CLINICAL TRIAL: NCT00431275
Title: An Open Label, Randomized Clinical Comparability Study Of The Current Liquid And Commercial Liquid Formulations
Brief Title: Study to Compare Two Formulations of CP-675,206 Monoclonal Antibody
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3671011
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commercial Formulation (Experimental): Commercial Formulation
  Interventions: Drug: CP-675,206
- Current Formulation (Experimental): Current Formulation
  Interventions: Drug: CP-675,206

INTERVENTIONS:
Drug: CP-675,206 — CP-675,206 15 mg/kg iv single dose on Day 1
  Other Names: anti-CTLA4 human monoclonal antibody
  Arms: Commercial Formulation
Drug: CP-675,206 — CP-675,206 15 mg/kg iv single dose on Day 1
  Arms: Current Formulation

SUMMARY:
This is an open-label, 2-arm study in which patients are randomized to receive either the formulation that is being used in clinical trials or the formulation that will be used when if the drug becomes commercially available. The purpose of this study is to compare the pharmacokinetics of the two formulations.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or Stage IV melanoma
* No evidence of disease following resection of melanoma lesions
* Recovered from all prior surgical or adjuvant treatment-related toxicities

Exclusion Criteria:

* History of chronic inflammatory or autoimmune disease
* History of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: maximum plasma concentration of CP-675,206 | 1 hour
Pharmacokinetics: AUC, defined as the area under the concentration -time curve | Time 0 to Day 85

SECONDARY OUTCOMES:
Human-anti-human antibodies | 1 year
Adverse events | 1 year
Safety laboratory tests | 1 year
Proportion of patients alive and free of disease at 1 year | 1 year

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, Scottsdale, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania